CLINICAL TRIAL: NCT04559555
Title: Managed Access Program (MAP) to Provide Access to Nilotinib, for Patients With Relapsed or Refractory Philadelphia Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia (ALL)
Brief Title: MAP to Provide Access to Nilotinib, for Patients With Relapsed or Refractory Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107A2412
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-05

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: Nilotinib; Acute lymphoblastic leukemia; ALL; Philadelphia chromosome positive; Ph+
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib

INTERVENTIONS:
Drug: Nilotinib — The compassionate use dose of nilotinib is 400 mg orally twice daily and should not be taken with food

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to nilotinib for eligible patients diagnosed with relapsed or refractory Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
Currently, preliminary responses of nilotinib monotherapy in adults with refractory or relapsed Ph+ ALL show limited clinical benefit in this population of patients with a high unmet medical need. Remissions induced by imatinib are of short duration and resistance to imatinib represents a major clinical challenge. The exact benefit and role of nilotinib in this leukemia remains to be determined and requires further analysis. Until further data is available patients with Ph+ ALL should be treated with nilotinib through the Individual Patient Program.. Studies to date indicate that nilotinib may provide clinical benefit to Ph+ ALL patients and may represent a novel treatment option for these patients.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be fulfilled for the provision of Managed Access and will vary depending on the stage of the product lifecycle:

* An independent request should be received from the Treating Physician (in some instances from Health Authorities, Institutions or Governments);
* The patient to be treated has a serious or life threatening disease or condition, and no comparable or satisfactory alternative therapy is available to monitor or treat the disease or condition;
* The patient is not eligible or able to enroll in a clinical trial;
* There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated;
* Provision of the investigational product will not interfere with the initiation, conduct or completion of a Novartis clinical trial or overall development program and
* Such access provision as described above is allowed as per local laws and regulations.

Exclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Male or Female patients age ≥ 18 years
2. WHO Performance Status of 0, 1 or 2
3. Relapsed or refractory Ph+ ALL
4. Imatinib (or dasatinib) must be discontinued at least 5 days prior to beginning therapy
5. Normal organ, electrolyte and marrow functions as described below:

   * Absolute Neutrophil Count (ANC) ≥ 1.0 x 1000000000/L
   * Platelets 50 x 1000000000/L
   * Potassium ≥ LLN (Lower limit of normal) or corrected to within normal limits with supplements prior to the first dose of nilotinib
   * Total calcium (corrected for serum albumin) ≥ LLN
   * Magnesium ≥ LLN or corrected to within normal limits with supplements prior to the first dose of nilotinib medication
   * AST and ALT ≤ 2.5 x ULN or ≤ 5.0 x UL:N if considered due to tumor
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum amylase and lipase ≤ 1.5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult